CLINICAL TRIAL: NCT05047640
Title: A Single-Blind, Randomized, Controlled Trial Comparing BNT162b2 vs JNJ-78436735 Vaccine as a Booster Dose After Completion of BNT162b2 Vaccine in Solid Organ Transplant Recipients
Brief Title: COVID-19 3rd Dose Vaccine in Transplant Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficulty in recruitment
Sponsor: Giselle Guerra (Other)
Responsible Party: Sponsor-Investigator, Giselle Guerra, Medical Director of Transplant Services, University of Miami
Organization: University of Miami (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20210641
Record Dates: First submitted 2021-09-13; First posted 2021-09-17 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Covid19
Keywords: transplant patients
MeSH Terms: conditions — COVID-19 | interventions — BNT162 Vaccine; Ad26COVS1

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BNT162b2 vaccine Group (Experimental): Participants in this arm will receive one booster dose of the BNT162b2.
  Interventions: Biological: BNT162b2 vaccine
- JNJ-78436735 vaccine Group (Experimental): Participants in this arm will receive one booster dose of the JNJ-78436735
  Interventions: Biological: JNJ-78436735 Vaccine

INTERVENTIONS:
Biological: BNT162b2 vaccine — Single dose of 0.3 mL BNT162b2 vaccine administered intramuscularly in the deltoid muscle
  Arms: BNT162b2 vaccine Group
Biological: JNJ-78436735 Vaccine — Single dose JNJ-78436735 Vaccine administered intramuscularly in the deltoid muscle
  Arms: JNJ-78436735 vaccine Group

SUMMARY:
The purpose of this study is to investigate the efficient vaccine type as a booster dose for Coronavirus Disease of 2019 (COVID-19) in solid organ transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age and older
* Patients who had received a solid organ (kidney, liver, lung, heart, and pancreas) transplant patient from living or deceased donors.
* Patients with active graft with at least one immunosuppressive medication
* Completed two doses of BNT162b2 vaccination at least 28 days ago

Exclusion Criteria:

* Patient with non-active graft
* Any significant side effect with previous COVID-19 vaccination
* Within 28 days of BNT162b2 vaccine completion
* Already received more than and equal to three doses of COVID-19 vaccination
* Previously received COVID-19 vaccine other than BNT162b2 vaccine
* Previously received monoclonal Antibody treatment that are specifically directed against the spike protein for Severe Acute Respiratory Syndrome (SARS) Coronavirus 2 (CoV)-2 such as Mab, Bamlanivimab, etesevimab, Casirivimab, imdevimab, Sotrovimab and/or any combination.
* Thrombocytopenia (if less than 50,000 per microliter 30 days prior vaccination)
* History of Capillary Leak Syndrome
* Adults unable to consent
* Individuals who are not yet adults (younger than 18 year old)
* Vulnerable patients (prisoners)
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2022-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giselle Guerra, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Natori Y, Martin E, Mattiazzi A, Arosemena L, Burke GW, Munagala MR, Manickavel S, Sota K, Pallikkuth S, Chen J, Bini J, Simkins J, Anjan S, Vianna RM, Guerra G. Post hoc analysis: 6 Months immunogenicity after third dose of BNT162b2 vs JNJ-78,436,735 after two doses of BNT162b2 vaccine in solid organ transplant recipients. Immunol Lett. 2025 Jun;273:106968. doi: 10.1016/j.imlet.2024.106968. Epub 2025 Jan 9. PMID 39798807
- [Derived] Natori Y, Martin E, Mattiazzi A, Arosemena L, Ortigosa-Goggins M, Shobana S, Roth D, Kupin WL, Burke GW, Ciancio G, Morsi M, Phancao A, Munagala MR, Butrous H, Manickavel S, Sinha N, Sota K, Pallikkuth S, Bini J, Simkins J, Anjan S, Vianna RM, Guerra G. A Pilot Single-Blinded, Randomized, Controlled Trial Comparing BNT162b2 vs. JNJ-78436735 Vaccine as the Third Dose After Two Doses of BNT162b2 Vaccine in Solid Organ Transplant Recipients. Transpl Int. 2023 Apr 5;36:10938. doi: 10.3389/ti.2023.10938. eCollection 2023. PMID 37091963

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BNT162b2 Vaccine Group | JNJ-78436735 Vaccine Group
Started | 30 | 28
Completed | 30 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BNT162b2 Vaccine Group | JNJ-78436735 Vaccine Group | Total
Number analyzed (Participants) | 30 | 28 | 58
Age, Continuous [Median (Full Range); unit: years] | 59.5 [27 to 76] | 54.5 [26 to 79] | 57.5 [26 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 21 | 17 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 14 | 22
  Not Hispanic or Latino | 22 | 14 | 36
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 14 | 8 | 22
  White | 16 | 19 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Tested Positive for IgG Antibodies to the Anti-spike Protein of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2)
Description: Anti-spike protein of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-COV-2) virus Immunoglobulin G (IgG) positivity rate will be assessed from serum blood samples
Time Frame: Up to 1 month (post booster vaccination)
Population: One patient on JNJ-78436735 vaccine group was not included in the analysis due to acquiring COVID-19 infection prior to the second blood draw.
Measure: Number; unit: percentage of participants
Arm/Group | BNT162b2 Vaccine Group | JNJ-78436735 Vaccine Group
Number analyzed (Participants) | 30 | 27
percentage of participants | 83.3 | 85.2

2. Secondary Outcome: Proportion of Participants With a Positive COVID-19 Test
Description: As assessed by medical records and or patient's report
Time Frame: Up to 1 month (post third dose)
Population: One patient on JNJ-78436735 vaccine group was not included in the analysis due to acquiring Coronavirus-19 (COVID-19) infection prior to the second blood draw.
Measure: Number; unit: proportion of participants
Arm/Group | BNT162b2 Vaccine Group | JNJ-78436735 Vaccine Group
Number analyzed (Participants) | 30 | 27
proportion of participants | 0 | 0

3. Secondary Outcome: Number of Participants With COVID-19 Symptom Severity as Measured by the WHO Scale
Description: World Health Organization (WHO) scale is scored between from 0 -10.
  0: Uninfected; non-viral Ribonucleic Acid (RNA) detected
  1. Asymptomatic; viral RNA detected
  2. Symptomatic; Independent
  3. Symptomatic; Assistance needed
  4. Hospitalized; No oxygen therapy
  5. Hospitalized; oxygen by mask or nasal prongs
  6. Hospitalized; oxygen by Non-invasive Ventilation (NIV) or High flow
  7. Intubation and Mechanical ventilation, partial pressure of oxygen (pO2) /fraction of inspired oxygen (FIO2) >=150 or oxygen saturation (SpO2) /FIO2>=200
  8. Mechanical ventilation, (pO2/FIO2<150 OR SpO2/FIO2<200) or vasopressors (norepinephrine >0.3 microg/kg/min)
  9. Mechanical ventilation, pO2/FIO2<150 and vasopressors (norepinephrine >0.3 microg/kg/min), or Dialysis or extracorporeal membrane oxygenation (ECMO)
  10. Dead
Time Frame: Up to 1 month (post third dose)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BNT162b2 Vaccine Group | JNJ-78436735 Vaccine Group
Number analyzed (Participants) | 30 | 27
Participants
  WHO score of 0 | 30 | 27
  WHO score of 1 | 0 | 0
  WHO score of 2 | 0 | 0
  WHO score of 3 | 0 | 0
  WHO score of 4 | 0 | 0
  WHO score of 5 | 0 | 0
  WHO score of 6 | 0 | 0
  WHO score of 7 | 0 | 0
  WHO score of 8 | 0 | 0
  WHO score of 9 | 0 | 0
  WHO score of 10 | 0 | 0

4. Secondary Outcome: Number of Participants With Vaccine-related Adverse Events
Description: Number of Participants with vaccine-related adverse events as collected by the study team.
Time Frame: Up to 7 days (post third dose)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BNT162b2 Vaccine Group | JNJ-78436735 Vaccine Group
Number analyzed (Participants) | 30 | 27
Participants
  Local Reaction | 9 | 6
  Systemic reaction | 7 | 5

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | BNT162b2 Vaccine Group | JNJ-78436735 Vaccine Group
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/28
Other Adverse Events (participants affected / at risk) | 13/30 | 20/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BNT162b2 Vaccine Group (N=30) | JNJ-78436735 Vaccine Group (N=28)
Arm pain (Injury, poisoning and procedural complications) | 8 (9) | 5 (5)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 6 (6)
Fatigue (General disorders) | 4 (4) | 3 (3)
Fever (General disorders) | 2 (2) | 2 (2)
Blurred Vision (Eye disorders) | 1 (1) | 0 (0)
Breast Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
COVID19 Infection (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Kidney Transplant Incision Abscess (Renal and urinary disorders) | 1 (1) | 0 (0)
Lactic Acidosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Poor Balance (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Post COVID Chronic Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Syncytial Virus Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Right Low Extremity Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Seborreic Keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Bacterial Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chills (Infections and infestations) | 0 (0) | 1 (1)
Chronic T-cell Mediated Rejection (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dizziness and Weakness (Nervous system disorders) | 0 (0) | 1 (1)
Elevated Creatinine (Renal and urinary disorders) | 0 (0) | 1 (1)
Essential Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Generalized Weakness (General disorders) | 0 (0) | 1 (1)
Hypovolemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leg Swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lower Extremities Edema (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Perinephric fluid collection (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pruritus/ eye redness (Eye disorders) | 0 (0) | 1 (1)
Sepsis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Transplant Renal Artery Stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Tremors (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-07): https://cdn.clinicaltrials.gov/large-docs/40/NCT05047640/Prot_SAP_000.pdf